CLINICAL TRIAL: NCT03290690
Title: A Prospective, Single-blind Evaluation of the Positive Predictive Value (PPV) of the MolecuLight i:X™ Imaging Device to Predict the Presence of Pseudomonas Aeruginosa in Chronic Wounds
Brief Title: Positive Predictive Value (PPV) of Pseudomonas Aeruginosa
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MolecuLight Inc. (Industry)
Collaborators: Scarborough Rouge Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 16-102
Record Dates: First submitted 2017-09-18; First posted 2017-09-25 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Wound; Chronic Leg Ulcer; Wound Contamination
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Subjects: All subjects in this study will have their wounds imaged and assessed in the following manner:
  Capture and save ST-image Capture and save FL-image Identify discrete locations of cyan (blue/green) fluorescent bacteria (FL_C) Acquire sample of tissue where cyan fluorescent bacteria are present (using curette method) Consent patient for inclusion in this study Note location of sample acquisition by annotating FL-image obtained in step 2 Send sample for microbiology analysis Note naming of microbiology sample on Case Report Form

SUMMARY:
This is a non-randomized, single-blind post market clinical follow-up study for which 65 patients will be imaged at Rouge Valley Centenary Hospital (Scarborough and Rouge Hospital) who present with a chronic wound and are receiving standard wound care treatment. The MolecuLight i:X imaging device will be used by the study clinician as an adjunctive tool in the assessment of the wound and will be used to guide the targeted sampling of a wound (with curettage scraping), as per current standard of care in the principal investigator's wound care clinic. The acquired tissue sample will then be analysed using conventional gold standard semi-quantitative culture methods to determine bacterial species present, also as per current standard of care in this clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients presenting with a chronic wound (wound duration > 4 weeks) e.g. diabetic foot ulcer, venous leg ulcer, pressure ulcer, or other acceptable aetiology
2. 18 years or older

Exclusion Criteria:

1. Treatment with an investigational drug within 1 month before study enrolment
2. Inability to consent to medical photography (i.e. inability to understand consent process)
3. Any contra-indication to routine wound care and/or monitoring
4. Prior participation of the patient in this study (for the same wound or a different wound).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be treated at the Scarborough and Rouge Hospital as per the standard of care, which includes use of the MolecuLight i:X imaging device and targeted sampling of regions with bacterial fluorescence for microbiological analysis. Patients will be identified as candidates and consented by the study's principle investigator. The images which would be acquired for this study are currently part of the routine clinical wound care assessment process in the principle investigator's wound care clinic. However, during study enrollment subjects will be given as much time as required for their understanding of the basic study, to understand that their participation is optional, to understand that they will receive standard of care wound treatment whether or not they choose to participate, and to have any potential questions addressed.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2017-08-04 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the ability of the MolecuLight i:X Imaging Device to predicting the presence of Pseudomonas aeruginosa in chronic wounds | 1 hour
  Primary endpoint: correlation of localized cyan fluorescence signals in device acquired images with microbiological samples indicating Pseudomonas aeruginosa

CONTACTS AND LOCATIONS:
Overall Officials: Rose Raizman, Principal Investigator — Scarborough Rouge Hospital
Locations (1):
- Scarborough and Rouge Hospital, Scarborough Village, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No